CLINICAL TRIAL: NCT04585321
Title: Comparative Bioavailability and Local Tolerability of Two Topical Diclofenac Plasters Applied Once and Twice a Day to Healthy Volunteers With a Repeat Dose Regimen
Brief Title: Comparative Bioavailability and Local Tolerability of Two Topical Diclofenac Plasters Applied Once and Twice a Day
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EQI7_17_01
Record Dates: First submitted 2020-03-02; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-02

CONDITIONS: Bioequivalence Study
MeSH Terms: interventions — Diclofenac; diclofenac hydroxyethylpyrrolidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-R (Other): Part 1 (QD) and part 2 (BID):
  Period 1: Test drug (T): Diclofenac Sodium 140mg Medicated Plaster EQI7, topical plaster.
  Period 2: Reference drug (R): Flector® topical plaster containing 180 mg of diclofenac hydroxyethylpyrrolidine equivalent to 140 mg of sodium diclofenac.
  Interventions: Drug: Diclofenac Sodium 140mg Medicated Plaster; Drug: Flector® topical plaster containing 180 mg of diclofenac hydroxyethylpyrrolidine equivalent to 140 mg of sodium diclofenac
- R-T (Other): Part 1 (QD) and part 2 (BID):
  Period 1: Reference drug (R): Flector® topical plaster containing 180 mg of diclofenac hydroxyethylpyrrolidine equivalent to 140 mg of sodium diclofenac.
  Period 2: Test drug (T): Diclofenac Sodium 140mg Medicated Plaster EQI7, topical plaster.
  Interventions: Drug: Diclofenac Sodium 140mg Medicated Plaster; Drug: Flector® topical plaster containing 180 mg of diclofenac hydroxyethylpyrrolidine equivalent to 140 mg of sodium diclofenac

INTERVENTIONS:
Drug: Diclofenac Sodium 140mg Medicated Plaster — Part 1: two seven-day study periods, separated by at least 7 days of wash-out. In the first period, a single plaster of Test Drug or Reference Drug will be applied on the back (lumbar region) for seven consecutive days. In the second period, a single plaster of the Reference Drug or Test Drug will be applied on the back (lumbar region) daily for seven consecutive days.
  Part 2: two seven-day study periods separated by at least 7 days of wash-out. In the first period, the Test Drug or Reference Drug plaster will be applied on the back (lumbar region) twice a day. In the second period, the Reference Drug or Test Drug plaster will be applied on the back (lumbar region) twice a day.
  Other Names: EQI7
Drug: Flector® topical plaster containing 180 mg of diclofenac hydroxyethylpyrrolidine equivalent to 140 mg of sodium diclofenac — Part 1: two seven-day study periods, separated by at least 7 days of wash-out. In the first period, a single plaster of Test Drug or Reference Drug will be applied on the back (lumbar region) for seven consecutive days. In the second period, a single plaster of the Reference Drug or Test Drug will be applied on the back (lumbar region) daily for seven consecutive days.
  Part 2: two seven-day study periods separated by at least 7 days of wash-out. In the first period, the Test Drug or Reference Drug plaster will be applied on the back (lumbar region) twice a day. In the second period, the Reference Drug or Test Drug plaster will be applied on the back (lumbar region) twice a day.
  Other Names: Flector

SUMMARY:
Study Objectives Primary To evaluate the average bioequivalence in healthy volunteers between medicinal product of Diclofenac Sodium 140mg Medicated Plaster EQI7 in comparison to the reference medicinal product Flector®, applied once and twice a day.

Secondary To evaluate pharmacokinetic profile on Day 1, adhesivity, local tolerability and safety of medicinal product Diclofenac Sodium 140mg Medicated Plaster EQI7 in healthy volunteers in comparison to the reference medicinal product Flector®, applied once and twice a day.

DETAILED DESCRIPTION:
Study Objectives Primary To evaluate the average bioequivalence in healthy volunteers between medicinal product of Diclofenac Sodium 140mg Medicated Plaster EQI7 in comparison to the reference medicinal product Flector®, both formulated as topical plasters applied once and twice a day.

Secondary To evaluate pharmacokinetic profile on Day 1, adhesivity, local tolerability and safety of medicinal product Diclofenac Sodium 140mg Medicated Plaster EQI7 in healthy volunteers in comparison to the reference medicinal product Flector®, both formulated as topical plasters applied once and twice a day.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, Caucasian/White aged between 18 and 55 years.
2. BMI between 19 and 29 kg/m² included
3. Normal or non-clinical significant findings on the physical examination
4. Normal or non-clinical significant finding on the laboratory evaluations. Laboratory values outside the normal range will be carefully evaluated by the clinical investigator. Subject showing safety laboratory values outside the normal range, but judged not clinically significant, may be allowed to enter the study. For sodium and potassium no values outside the normal range will be allowed.
5. Willing and able to understand and sign an approved Informed Consent form.
6. If female, they must not be pregnant or breast feeding and using an effective contraception method during the study (hormonal, such as birth control pill, or barrier method, such as condom or diaphragm, or intrauterine, such as spiral).

Exclusion Criteria:

1. History of alcohol or drug abuse.
2. Smokers of more than 10 cigarettes/day.
3. History of gastrointestinal, renal, hepatic, pulmonary or cardiovascular disease; or history of epilepsy, asthma, diabetes, psychosis or glaucoma.
4. History of allergic response to diclofenac or related drugs, namely non-steroidal anti-inflammatory agents
5. Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis)
6. Participation in a previous clinical trial within the past 6 months.
7. Blood donation of 250 ml or more within the past 3 months.
8. Treatment with any known enzyme inhibiting or inducing agents (barbiturates, phenothiazines, etc.) within the past 4 weeks.
9. Positive to HIV test and/or Hepatitis B and C tests.
10. Positive to drugs of abuse qualitative screen in urine.
11. Use of any prescription or over-the-counter medication on a regular basis.
12. Drinking excessive amounts of tea, cacao, coffee and/or beverages containing caffeine (> 5 cups/day) or wine (> 0,5 l/day) or spirits (> 50 ml/day)
13. In the judgement of the Clinical Investigator subjects likely to be not compliant or cooperative during the study.
14. Irritation scale score higher than zero at the sites of application.
15. Presence of skin injuries at the sites of application.
16. An acquired tan (by sun or lamp) in the previous 2 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Css max (ng/mL) of Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 7 through Day 9 | Day 7 through Day 9
  Css max on Day 7 through Day 9
AUCττ (ng/mL*h) of Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 7 through Day 9 | Day 7 through Day 9
  AUCττ on Day 7 through Day 9

SECONDARY OUTCOMES:
Cmax (ng/mL) of Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 | Day 1
  Cmax on Day 1
AUC (ng/mL*h) of Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 | Day 1
  AUC on Day 1
Adhesivity of Diclofenac Sodium 140mg Medicated Plaster EQI7 in comparison to Flector® topical plasters applied once and twice a day with a 5-point ordinal scale, where 0= >90%adhered and 4=plaster detached, from Day 1 for the entire study period | From Day 1 for the entire study duration
  Adhesivity of plasters with adhesivity 5-point ordinal scale:
  0 = >90% adhered; 1 = >75% to <90% adhered; 2 = >50% to <75% adhered; 3 =< 50% adhered but not detached; 4 = Plaster detached, from Day 1 for the entire study period
Local tolerability of Diclofenac Sodium 140mg Medicated Plaster EQI7 in comparison to Flector® topical plasters applied once and twice a day, with the irritation8-point scale, where 0=no evidence of irritation and 7=strong reaction, from Day1 onward | From Day 1 for the entire study duration
  Local tolerability: irritation 8-point categorical scale:0=no evidence of irritation;1=minimal erythema, barely perceptible;2=definite erythema, readily visible;3=minimal edema or minimal papular response;3=erythema and papules;4=definite edema;5=erythema, edema, and papules;6=vescicular eruption;7=strong reaction spreading beyond test site, from Day1 for the entire study duration
Local tolerability of Diclofenac Sodium 140mg Medicated Plaster EQI7 in comparison to Flector® topical plasters applied once and twice a day, with the syntoms 4-point categorical scale score, where 0=absent and 3=severe, from Day1 onward | From Day 1 for the entire study duration
  Local tolerability: symptoms 4-point categorical scale:0=absent;1=mild;2=moderate;3=severe), from Day1 for the entire study duration
Measurement of heart rate in bpm during treatment with Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 of period 1 and Day 9 of period 2 | Day 1 of period 1 and Day 9 of period 2
  Heart rate measurement in bpm on Day 1 of period 1 and Day 9 of period 2
Measurement of systolic/diastolic blood pressure in mmHg during treatment with Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 of period 1 and Day 9 of period 2 | Day 1 of period 1 and Day 9 of period 2
  Systolic/diastolic blood pressure in mmHg measurement on Day 1 of period 1 and Day 9 of period 2
Measurement of body temperature in C degree during treatment with Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 of period 1 and Day 9 of period 2 | Day 1 of period 1 and Day 9 of period 2
  Body temperature in C degrees measurement on Day 1 of period 1 and Day 9 of period 2
Haematological analysis during treatment with Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 of period 1 and Day 9 of period 2 | Day 1 of period 1 and Day 9 of period 2
  Haematological analysis on Day 1 of period 1 and Day 9 of period 2
Biochemical analysis during treatment with Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 of period 1 and Day 9 of period 2 | Day 1 of period 1 and Day 9 of period 2
  Biochemical analysis on Day 1 of period 1 and Day 9 of period 2
Virological tests during treatment with Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 of period 1 and Day 9 of period 2 | Day 1 of period 1 and Day 9 of period 2
  Virological tests on Day 1 of period 1 and Day 9 of period 2
Urinalysis during treatment with Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 of period 1 and Day 9 of period 2 | Day 1 of period 1 and Day 9 of period 2
  Urinalysis on Day 1 of period 1 and Day 9 of period 2
12-lead ECG evaluation during treatment with Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day on Day 1 of period 1 and Day 9 of period 2 | Day 1 of period 1 and Day 9 of period 2
  12-lead ECG on Day 1 of period 1 and Day 9 of period 2
Incidence of adverse events using Diclofenac Sodium 140mg Medicated Plaster EQI7 and Flector® topical plasters applied once and twice a day from Day 1 for the entire study duration | From Day 1 for the entire study duration
  Incidence of adverse events from Day 1 for the entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Giordan, Study Director — Fidia Farmaceutici s.p.a.
Locations (1):
- CRC Centro Ricerche Cliniche di Verona s.r.l. c/o Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No